CLINICAL TRIAL: NCT05354661
Title: Non-Invasive Hemodynamic Monitoring and Incidence of Perioperative Hypotension in Gynaecologic Oncologic Surgery: Hypotension Prediction Index Working With ClearSight Versus Arterial Waveform Analysis Alone
Brief Title: Perioperative Hypotension in Gynaecologic Oncologic Surgery: HPI-ClearSight Versus Arterial Waveform Analysis
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3664
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-04

CONDITIONS: Hypotension; Hemodynamic Instability; Gynecologic Cancer
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypotension Prediction Index (HPI) group: Hemodinamic monitoring with HPI working with ClearSight
  Interventions: Device: Hypotension Prediction Index
- Control group: Hemodinamic monitoring with classic ClearSight

INTERVENTIONS:
Device: Hypotension Prediction Index — treatment of hypotension before the appearance following HPI algorithm
  Groups: Hypotension Prediction Index (HPI) group

SUMMARY:
Background Intraoperative hypotension is associated with increased morbidity and mortality. The Hypotension Prediction Index (HPI) is an advancement of the arterial waveform analysis to predict intraoperative hypotension minutes before episodes occur enabling preventive treatments.

This study will test the hypothesis that a hemodynamic treatment protocol based on HPI working with non-invasive ClearSight system reduces intraoperative hypotension when compared to standard goal directed therapy (GDT) in patients undergoing gynaecologic oncologic surgery.

Methods A retrospective analysis of 68 adult consecutive patients undergoing gynaecologic oncologic surgery with non-invasive arterial pressure monitoring using either index guidance (HPI) or classic ClearSight system waveform analysis depending on availability (ClearSight, n = 36; HPI, n = 32) will be conducted. A hemodynamic GDT protocol was applied in both groups. The primary endpoint will be the incidence and duration of hypotensive events defined as MAP <65 mmHg evaluated by time-weighted average of hypotension.

DETAILED DESCRIPTION:
INTRODUCTION Intraoperative hypotension (IOH) is a common adverse event during noncardiac surgery [1,2]. It is associated with an increased incidence of acute kidney injury, myocardial injury, neurological deficiencies, as well as an increased 30-day operative mortality [3-7]. Organ injuries were shown to be associated with the depth, frequency, and duration of hypotensive episodes [4,8]. Data indicate that a mean arterial pressure of 65 mmHg serves as a threshold to predict myocardial and kidney injury [9-11].

Recently developed minimally invasive methods of the arterial waveform analysis allow calculation of cardiac output, stroke volume, stroke volume variation, and systemic vascular resistance. This deeper insight into hemodynamics enables goal-directed therapy approaches; however, the given information only allows to react to events instead of preventing them [12,13].

Interestingly, recent data indicate a significant reduction in postoperative organ dysfunction by preventing IOH, suggesting a potential benefit of early intervention [14].

Surgical interventions for cancer mass reduction are among the most invasive operations in gynaecology. Extensive surgical trauma results in severe intra- and perioperative volume shifts and unstable hemodynamics [15]. Major abdomino-pelvic surgery for gynaecological oncologic surgery (GOS) may include hysterectomy, oophorectomy, omentectomy, colectomy, removal of the lymph nodes and peritoneal stripping. Surgery is carried out through laparoscopy or a laparotomic incision and is often associated with significant blood loss [16]. Hypotension during GOS is common, and as it is associated with the potential for harm, it requires prompt evaluation and treatment [16]. Extensive fluid resuscitation in peritoneal cancer patients is associated with a poor postoperative outcome independent from the underlying malignant disease and avoiding fluid overload is recommended [15].

Therefore, the prediction of intraoperative hypotension and consequently its prevention by proactive treatment may show beneficial effects for patients. Machine learning, a discipline within computer science used to analyse large data sets and to develop predictive models, has evident applications in health care [17,18]. Several attempts to use algorithms as an aid in anaesthesiology practice recently received renewed attention, with the aim of optimizing patients' perioperative status, primarily focusing on detection of early hemodynamic instability and prediction of hypotension [19].

The Hypotension Prediction Index - HPI (Edwards Lifesciences, Irvine, USA) is an algorithm based on the complex analysis of features in high fidelity arterial pressure waveform recordings developed to observe subtle signs that could predict the onset of hypotension in surgical and intensive care unit patients [20]. HPI is a unitless number that ranges from 1 to 100, and as the number increases, the likelihood or risk of a hypotensive event (defined as a mean arterial pressure [MAP] <65 mmHg for more than 1 minute) occurring in the near future increases [20]. A validation study conducted on surgical patients reported high sensitivity and specificity of HPI for predicting hypotension 5, 10 and 15 min before the event occurred [21]. The development of the algorithm was based on invasive arterial line waveform data; however, only a small fraction of patients having noncardiac surgery requires invasive arterial monitoring [22].

Estimation of arterial pressure waveforms from a non-invasive finger cuff (ClearSight) is well established, and MAP measured by ClearSight system could be considered as an alternative for mean radial arterial pressure [23,24]. The HPI algorithm, is recently reported to work also with a non-invasive waveform estimate [25-27].

This study will compare a hemodynamic management based on the HPI algorithm working with non-invasive ClearSight system with a classic ClearSight-based one in terms of incidence, duration, and severity of intraoperative hypotensive events evaluated by time-weighted average of hypotension in patients undergoing GOS.

MATERIALS AND METHODS This single-center retrospective observational study was approved by the Internal Ethics Committee (ID 3664, protocol number 10077/21). Written informed consent will be obtained from all the patients involved.

The primary endpoint is the incidence, duration, and severity of hypotensive events (defined as MAP < 65 mmHg for at least 1 minute) evaluated by time-weighted average (TWA) MAP of hypotension in the two groups of patients. The TWA-MAP is a combination of severity and duration of the hypotensive events, in relation to the total surgery time. It is calculated by using the sum of the area under the threshold divided by the duration of surgery [28]. The threshold for hypotensive events is defined as a MAP below 65 mmHg for at least 1-min duration. Hypotension duration time ends after re-increasing MAP values upon ≥65 mmHg for at least 1 min.

Secondary endpoints consists of number of patients with hypotensive events, number of events per (respective) patient, cumulative and average duration of hypotension, combined with numbers of hypotensive events <65 and <50 mmHg.

The data were collected during a limited period of time in which new hemodynamic monitoring sensors (ClearSight) were evaluated during a time marketing release. The first 68 patients undergoing GOS at IRCCS Policlinico A.Gemelli Foundation between December 2019 and February 2020 were monitored either with classic ClearSight sensor (n= 36) and ClearSight sensor with HPI-enabled (n = 32). Inclusion criteria consisted of elective GOS, age >18 years. Exclusion criteria were patients not in sinus rhythm, ejection fraction <30%, severe aortic valve stenosis, emergency surgery, acute myocardial ischemia, pregnancy.

Standard monitoring (Life Scope TR, Nihon Kohden Co, Tokyo, Japan) included a 5-lead electrocardiogram, pulse oximetry, non-invasive blood pressure (NIBP) and eventual invasive blood pressure (IBP). In addition to standard monitoring, all patients had a non-invasive hemodynamic monitoring with ClearSight (Edwards Lifesciences, Irvine, CA). After arriving at the operating theatre, NIBP measurement using an automated digital sphygmomanometer on the right arm was started and the ClearSight system was attached to a finger of the left arm of the patients. We connected the ClearSight monitor with an interface cable to the patient monitor. In patients requiring IBP monitoring an arterial cannula was placed contralateral to the ClearSight cuff. The ClearSight reference system was zeroed at the level of the right atrium. The blood pressure value from the finger cuff (CS-BP) was reported on the main monitor. NIBP measurement using the automated digital sphygmomanometer was performed at 5-min intervals. For therapy purposes we defined hypotension as an absolute value of CS-BP MAP < 65 mmHg. Incidence and duration of hypotensive episodes and interventions were registered. Bradycardia was defined as a heart rate (HR) < 60 bpm.

A large bore i.v. catheter was inserted in a forearm vein, and Cefazoline 2 gr, Dexamethasone 4 mg and Omeprazole 40 mg were administered. General anesthesia was induced with sufentanil 0.2 mcg/kg (ideal body weight), propofol 2 mg/kg (actual body weight), and rocuronium 0.6 mg/kg (ideal body weight). During surgery, patients were positioned in Trendelenburg position with both arms spread out on arm-positioning devices. Anesthesia was maintained with Sevoflurane to maintain a Bispectral Index value between 40-50. Additional boluses of sufentanil and rocuronium were administered when needed.

All patients received a GDT hemodynamic protocol to optimize the cardiac output and oxygen supply. As part of the GDT protocol, patients received crystalloid and/or fluids to maintain SVV<13% or to avoid SV decrease of more than 10% of the baseline. Vasopressor and inotropic medication were administered upon request of the clinician in order to maintain a MAP ≥65. In the HPI group, the attending anesthesiologist was free to use liquid, vasopressors and inotropic drugs, but he was allowed to read on the Hemosphere monitor HPI and secondary parameters (for evaluation of preload, cardiac contractility, and afterload as possible causes for hypotension), and to act in a preventive way in order to avoid hypotension.

All data were downloaded from the HemoSphere monitor, including HPI, CS-MAP, CS systolic arterial pressure, CS diastolic arterial pressure. All downloaded data consisted of 20-second interval averaged data points. Data were transferred to a computer for analysis via an USB drive. Every file was appointed with an automated generated code by the machine and was identifiable by an ID number contained within it.

The HPI algorithm estimates the probability of occurrence in the near future of a hypotensive event taking the arterial pressure waveform as the input to compute an index value that ranges between 1 and 100. In this study, instead of invasive arterial waveform data, we used the non-invasive arterial pressure waveform of ClearSight.

In the HemoSphere monitor, poor quality arterial waveforms were automatically detected by the arterial waveform processing algorithms and excluded from the computation of the 20-sec averages.

Statistical analysis Data collected perioperatively and downloaded from the HemoSphere platform will be analyzed using the Acumen Analytics Software (Edwards Lifesciences Corp.).

Categorical data will be presented as frequencies with percentages. Differences will be analyzed with the Fisher's exact test. For quantitative variables test for normal distribution with the Shapiro-Wilk test will be used. Data will be presented as means ±standard deviation (SD) in case of normally distribution, otherwise, as median and interquartile range (IQR). Linear variables will be analyzed using the Student's unpaired t-test in normal distributed variables and the Mann-Whitney U-test in non-normally distributed variables. P-values less than 0.05 will be considered statistically significant. Statistical analysis will be performed with SPSS Statistics.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic Oncologic surgery procedures

Exclusion Criteria:

* Severe valvulopathy
* Cardiac failure
* Severe aortic stenosis
* Severe cardiac arrhythmias
* Coagulopathy
* Contraindication to arterial calculation
* Patient's refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent gynaecologic oncologic surgery between december 2019 and february 2020
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Cumulative Intraoperative Hypotension | At the end of surgery
  Comparison, in the two groups, of the amount of intraoperative hypotension (MAP < 65 mmHg), measured with TWAMAP method.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bijker JB, van Klei WA, Kappen TH, van Wolfswinkel L, Moons KG, Kalkman CJ. Incidence of intraoperative hypotension as a function of the chosen definition: literature definitions applied to a retrospective cohort using automated data collection. Anesthesiology. 2007 Aug;107(2):213-20. doi: 10.1097/01.anes.0000270724.40897.8e. PMID 17667564
- [Result] Vernooij LM, van Klei WA, Machina M, Pasma W, Beattie WS, Peelen LM. Different methods of modelling intraoperative hypotension and their association with postoperative complications in patients undergoing non-cardiac surgery. Br J Anaesth. 2018 May;120(5):1080-1089. doi: 10.1016/j.bja.2018.01.033. Epub 2018 Mar 21. PMID 29661385
- [Result] An R, Pang QY, Liu HL. Association of intra-operative hypotension with acute kidney injury, myocardial injury and mortality in non-cardiac surgery: A meta-analysis. Int J Clin Pract. 2019 Oct;73(10):e13394. doi: 10.1111/ijcp.13394. Epub 2019 Sep 11. PMID 31332896
- [Result] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Result] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Result] Scholz AF, Oldroyd C, McCarthy K, Quinn TJ, Hewitt J. Systematic review and meta-analysis of risk factors for postoperative delirium among older patients undergoing gastrointestinal surgery. Br J Surg. 2016 Jan;103(2):e21-8. doi: 10.1002/bjs.10062. Epub 2015 Dec 16. PMID 26676760
- [Result] Bijker JB, Persoon S, Peelen LM, Moons KG, Kalkman CJ, Kappelle LJ, van Klei WA. Intraoperative hypotension and perioperative ischemic stroke after general surgery: a nested case-control study. Anesthesiology. 2012 Mar;116(3):658-64. doi: 10.1097/ALN.0b013e3182472320. PMID 22277949
- [Result] Ahuja S, Mascha EJ, Yang D, Maheshwari K, Cohen B, Khanna AK, Ruetzler K, Turan A, Sessler DI. Associations of Intraoperative Radial Arterial Systolic, Diastolic, Mean, and Pulse Pressures with Myocardial and Acute Kidney Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2020 Feb;132(2):291-306. doi: 10.1097/ALN.0000000000003048. PMID 31939844
- [Result] Mascha EJ, Yang D, Weiss S, Sessler DI. Intraoperative Mean Arterial Pressure Variability and 30-day Mortality in Patients Having Noncardiac Surgery. Anesthesiology. 2015 Jul;123(1):79-91. doi: 10.1097/ALN.0000000000000686. PMID 25929547
- [Result] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Result] Mathis MR, Naik BI, Freundlich RE, Shanks AM, Heung M, Kim M, Burns ML, Colquhoun DA, Rangrass G, Janda A, Engoren MC, Saager L, Tremper KK, Kheterpal S, Aziz MF, Coffman T, Durieux ME, Levy WJ, Schonberger RB, Soto R, Wilczak J, Berman MF, Berris J, Biggs DA, Coles P, Craft RM, Cummings KC, Ellis TA 2nd, Fleishut PM, Helsten DL, Jameson LC, van Klei WA, Kooij F, LaGorio J, Lins S, Miller SA, Molina S, Nair B, Paganelli WC, Peterson W, Tom S, Wanderer JP, Wedeven C; Multicenter Perioperative Outcomes Group Investigators. Preoperative Risk and the Association between Hypotension and Postoperative Acute Kidney Injury. Anesthesiology. 2020 Mar;132(3):461-475. doi: 10.1097/ALN.0000000000003063. PMID 31794513
- [Result] Suehiro K, Tanaka K, Mikawa M, Uchihara Y, Matsuyama T, Matsuura T, Funao T, Yamada T, Mori T, Nishikawa K. Improved Performance of the Fourth-Generation FloTrac/Vigileo System for Tracking Cardiac Output Changes. J Cardiothorac Vasc Anesth. 2015;29(3):656-62. doi: 10.1053/j.jvca.2014.07.022. Epub 2014 Nov 14. PMID 25440654
- [Result] Kouz K, Scheeren TWL, de Backer D, Saugel B. Pulse Wave Analysis to Estimate Cardiac Output. Anesthesiology. 2021 Jan 1;134(1):119-126. doi: 10.1097/ALN.0000000000003553. No abstract available. PMID 32914174
- [Result] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Result] Gehlen J, Klaschik S, Neumann C, Keyver-Paik MD, Mustea A, Soehle M, Frede S, Velten M, Hoeft A, Hilbert T. Dynamic changes of angiopoietins and endothelial nitric oxide supply during fluid resuscitation for major gyn-oncological surgery: a prospective observation. J Transl Med. 2020 Jan 31;18(1):48. doi: 10.1186/s12967-020-02236-9. PMID 32005259
- [Result] Bossy M, Nyman M, Madhuri TK, Tailor A, Chatterjee J, Butler-Manuel S, Ellis P, Feldheiser A, Creagh-Brown B. The need for post-operative vasopressor infusions after major gynae-oncologic surgery within an ERAS (Enhanced Recovery After Surgery) pathway. Perioper Med (Lond). 2020 Sep 7;9:26. doi: 10.1186/s13741-020-00158-0. eCollection 2020. PMID 32939254
- [Result] Frizzell JD, Liang L, Schulte PJ, Yancy CW, Heidenreich PA, Hernandez AF, Bhatt DL, Fonarow GC, Laskey WK. Prediction of 30-Day All-Cause Readmissions in Patients Hospitalized for Heart Failure: Comparison of Machine Learning and Other Statistical Approaches. JAMA Cardiol. 2017 Feb 1;2(2):204-209. doi: 10.1001/jamacardio.2016.3956. PMID 27784047
- [Result] Pinsky MR. Complexity modeling: identify instability early. Crit Care Med. 2010 Oct;38(10 Suppl):S649-55. doi: 10.1097/CCM.0b013e3181f24484. PMID 21164410
- [Result] Guillame-Bert M, Dubrawski A, Wang D, Hravnak M, Clermont G, Pinsky MR. Learning temporal rules to forecast instability in continuously monitored patients. J Am Med Inform Assoc. 2017 Jan;24(1):47-53. doi: 10.1093/jamia/ocw048. Epub 2016 Jun 6. PMID 27274020
- [Result] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Result] Davies SJ, Vistisen ST, Jian Z, Hatib F, Scheeren TWL. Ability of an Arterial Waveform Analysis-Derived Hypotension Prediction Index to Predict Future Hypotensive Events in Surgical Patients. Anesth Analg. 2020 Feb;130(2):352-359. doi: 10.1213/ANE.0000000000004121. PMID 30896602
- [Result] Nuttall G, Burckhardt J, Hadley A, Kane S, Kor D, Marienau MS, Schroeder DR, Handlogten K, Wilson G, Oliver WC. Surgical and Patient Risk Factors for Severe Arterial Line Complications in Adults. Anesthesiology. 2016 Mar;124(3):590-7. doi: 10.1097/ALN.0000000000000967. PMID 26640979
- [Result] Ameloot K, Palmers PJ, Malbrain ML. The accuracy of noninvasive cardiac output and pressure measurements with finger cuff: a concise review. Curr Opin Crit Care. 2015 Jun;21(3):232-9. doi: 10.1097/MCC.0000000000000198. PMID 25922896
- [Result] Saugel B, Hoppe P, Nicklas JY, Kouz K, Korner A, Hempel JC, Vos JJ, Schon G, Scheeren TWL. Continuous noninvasive pulse wave analysis using finger cuff technologies for arterial blood pressure and cardiac output monitoring in perioperative and intensive care medicine: a systematic review and meta-analysis. Br J Anaesth. 2020 Jul;125(1):25-37. doi: 10.1016/j.bja.2020.03.013. Epub 2020 May 29. PMID 32475686
- [Result] Maheshwari K, Buddi S, Jian Z, Settels J, Shimada T, Cohen B, Sessler DI, Hatib F. Performance of the Hypotension Prediction Index with non-invasive arterial pressure waveforms in non-cardiac surgical patients. J Clin Monit Comput. 2021 Feb;35(1):71-78. doi: 10.1007/s10877-020-00463-5. Epub 2020 Jan 27. PMID 31989416
- [Result] Wijnberge M, van der Ster BJP, Geerts BF, de Beer F, Beurskens C, Emal D, Hollmann MW, Vlaar APJ, Veelo DP. Clinical performance of a machine-learning algorithm to predict intra-operative hypotension with noninvasive arterial pressure waveforms: A cohort study. Eur J Anaesthesiol. 2021 Jun 1;38(6):609-615. doi: 10.1097/EJA.0000000000001521. PMID 33927105
- [Result] Frassanito L, Giuri PP, Vassalli F, Piersanti A, Longo A, Zanfini BA, Catarci S, Fagotti A, Scambia G, Draisci G. Hypotension Prediction Index with non-invasive continuous arterial pressure waveforms (ClearSight): clinical performance in Gynaecologic Oncologic Surgery. J Clin Monit Comput. 2022 Oct;36(5):1325-1332. doi: 10.1007/s10877-021-00763-4. Epub 2021 Oct 7. PMID 34618291
- [Result] Maheshwari K, Khanna S, Bajracharya GR, Makarova N, Riter Q, Raza S, Cywinski JB, Argalious M, Kurz A, Sessler DI. A Randomized Trial of Continuous Noninvasive Blood Pressure Monitoring During Noncardiac Surgery. Anesth Analg. 2018 Aug;127(2):424-431. doi: 10.1213/ANE.0000000000003482. PMID 29916861